CLINICAL TRIAL: NCT01317134
Title: Serological and Non-invasive Evaluation of Endothelial Function in Patients With Pulmonary Arterial Hypertension
Brief Title: Endothelial Function in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Pfizer (Industry); Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PNEU-PV3334/2009/UKE
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Pathophysiology; Genetics
Keywords: Pulmonary Arterial Hypertension; Prognostic factors; Signal transduction; Genetics
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Therapy-naive (Active Comparator): This group consists of patients with a newly diagnosed PH (Class I or IV). First blood sampling takes place before initiation of PH therapy (0 months), the following measurements will be performed after 3, 6, 9 and 12 months under specific therapy.
  Initiation of standard therapy is performed directly after baseline visit / study inclusion. No special study medication will be used.
  Intervention: a) Device: EndoPAT measurement and b) Biological/Vaccine: Blood Test
  Interventions: Device: EndoPAT measurement; Biological: Blood Test
- Under therapy (Active Comparator): This group consists of patients under ERA monotherapy at timepoint of inclusion. Observation period is one year to detect intraindividual changes in endothelial dysfunction measured by L-arginine/NO-metabolites after 0, 3, 6, 9 and 12 months under investigation.
  Specific PAH therapy has been started prior to the study for medical reasons and will be continued throughout.
  Intervention: a) Device: EndoPAT measurement and b) Biological/Vaccine: Blood
  Interventions: Device: EndoPAT measurement; Biological: Blood Test
- Healthy controls (Active Comparator): This group consists of healthy individuals. Sex and age matching is intended. Intervention: a) Device: EndoPAT measurement and b) Biological/Vaccine: Blood
  Interventions: Device: EndoPAT measurement; Biological: Blood Test

INTERVENTIONS:
Device: EndoPAT measurement — EndoPAT (Itamar Medical Ltd, Ceasarea, Isreal) quantifies the endothelium-mediated changes in vascular tone, elicited by a 5-minute occlusion of the brachial artery (using a standard blood pressure cuff). When the cuff is released, the surge of blood flow causes an endothelium-dependent Flow Mediated Dilatation (FMD). The dilatation, manifested as Reactive Hyperemia, is captured by EndoPAT as an increase in the PAT Signal amplitude. A post-occlusion to pre-occlusion ratio is calculated by the EndoPAT software, providing the EndoPAT index. EndoPAT is FDA-cleared and CE-marked.
Biological: Blood Test — It is hypothesized that L-arginine/NO-metabolites are altered in pulmonary hypertension depending on disease severity. Moreover, polymorphisms in L-arginine/NO-metabolism modifying factors may influence disease severity. Analysis will be performed following established/published protocols after isolation from whole blood.

SUMMARY:
The objectives of the current study are to identify and evaluate new prognostic non-invasive and serological markers in patients with pulmonary hypertension. The focus will be on L-arginine metabolism and to clarify its influence on endothelial function.

DETAILED DESCRIPTION:
The objectives of the current study are to identify and evaluate new prognostic non-invasive and serological markers in patients with pulmonary hypertension. The focus will be on L-arginine metabolism and to clarify its influence on endothelial function. The investigators also want to evaluate differences in plasma concentrations of L-arginine/NO metabolites and non-invasively assessed endothelial function based on specific PH-therapy.

Furthermore, the investigators aim to transfer the results gained from the investigators study population to in-vitro systems in order to carefully characterize the involved signal transduction pathways. Thereby the investigators hope to identify potentially new therapeutic targets in PH or patient subgroups preferably benefitting from established therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* proven PH (by right heart catheterization, PAP >25 mmHg, within last 12 months)
* age >18 years
* Dana Point classification I or IV (all subgroups)
* declaration of consent

Exclusion Criteria:

* Pulmonary Hypertension not proven by right heart catheterization
* Eisenmenger's syndrome/reaction
* PH other than Dana Point I and IV
* alcohol or drug abuse
* non-compliance due to any cause (e.g. severe psychiatric disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Differences of endothelial function regarding disease class and severity | 0, 3, 6, 9 and 12 months
  1. Quantification of L-arginine metabolites in whole blood
  2. PAT-Ratio as non-invasively assessed endothelial function by EndoPAT2000-Device (Itamar Medical Ltd., Caesarea, Israel)
  0 months = Time of Inclusion

SECONDARY OUTCOMES:
Correlation of endothelial function with changes in pulmonary hemodynamics | 0,3,6,9 and 12 months
  L-arginine metabolite concentrations and PAT-Ratio correlated with PAPm, RAP, PVR (assessed by right heart catheterization within 12 months prior to inclusion) and echocardiographical parameters RVSP, TAPSE and TEI.
Correlation of endothelial function with established prognostic factors | 0,3,6,9 and 12 months
  L-arginine metabolite concentrations and PAT-Ratio correlated with plasma concentration of proBNP as well as capillary pCO2, 6-minute walk distance and NYHA/WHO functional class.
Correlation of endothelial function with possible prognostic factors | 0,3,6,9 and 12 months
  L-arginine metabolite concentrations and PAT-Ratio correlated with plasma concentration of various enzymes as well as lung function.
Correlation of L-arginine metabolites with pulmonary vascular signaling | 0 months
  In vitro evaluation of human pulmonary vasculature cells signaling and proliferation by altered L-arginine metabolite levels.
Correlation of polymorphisms in L-arginine metabolism genes with disease severity | 0 months
Correlation of endothelial function with possible novel diagnostic or prognostic factors (e.g., inflammatory markers, intermediary metabolites) | 0 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans FE Klose, MD, Study Director — Department of Respiratory Medicine, University Medical Center Hamburg-Eppendorf; Jan K Hennigs, MD, Principal Investigator — Department of Respiratory Medicine, University Medical Center Hamburg - Eppendorf
Locations (1):
- Department of Respiratory Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to Publication of Study Results — https://ediss.sub.uni-hamburg.de/handle/ediss/7300